CLINICAL TRIAL: NCT04571489
Title: Gimatecan (ST1481) as Second-line Treatment for Locally Advanced or Metastatic Pancreatic Cancer: an Open-label, Randomized, Controlled Phase II Study
Brief Title: A Phase II Study of Gimatecan (ST1481) in Locally Advanced or Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST1481-LEES-2020-05
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; chemotherapy; gimatecan
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ST 1481; Tegafur; gimeracil; potassium oxonate; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gimatecan group (Experimental): All patients will receive gimatecan (0.8mg/m2, on days 1 to 5, PO, every 4 weeks) until progressive disease (PD).
  Interventions: Drug: Gimatecan
- placebo group (Placebo Comparator): All patients will receive tegafur, gimeracil and oteracil potassium (40-60mg, twice daily, on days 1 to 14 , PO, every 3 weeks) or gemcitabine (1000mg/m2, on days 1、8, IV, every 3 weeks) until progressive disease (PD).
  Interventions: Drug: tegafur, gimeracil and oteracil potassium; Drug: gemcitabine

INTERVENTIONS:
Drug: Gimatecan — Patients will receive gimatecan orally at 0.8mg/m2 on day 1-5 every 4 weeks.
  Other Names: ST1481
  Arms: Gimatecan group
Drug: tegafur, gimeracil and oteracil potassium — Patients will receive tegafur, gimeracil and oteracil potassium orally at 40 or 60mg twice daily on days 1 to 14 every 3 weeks.
  Arms: placebo group
Drug: gemcitabine — Patients will receive gemcitabine IV at 1000mg/m2 on days 1、8 every 3 weeks.
  Arms: placebo group

SUMMARY:
This phase II clinical trial studies the safety and effect of as second-line treatmen in local advanced or metastatic pancreatic cancer. The Gimatecan will be given every four weeks.

ELIGIBILITY:
Key inclusion Criteria:

1. Histologically or cytologically confirmed pancreatic cancer originating from pancreatic ductal epithelium, excluding pancreatic endocrine tumor;
2. Locally advanced or metastatic pancreatic cancer in no condition for radical radiotherapy or operation;
3. Failed in first-line gemcitabine or fluorouracil drugs chemotherapy (Recurrence within 6 months after treatment, progression or toxicity intolerance during treatment);
4. Chemotherapy, targeted therapy or radical radiotherapy should be stopped 3 weeks ago, immunotherapy should be stopped 4 weeks ago, and previous toxicity recovered (CTCAE ≤ level 1);
5. Measurable cancer lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
6. No younger than 18 years old of either gender;
7. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1;
8. Estimated life expectancy >3 months;
9. The function of important organs meets the following requirements:

   1. absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets ≥ 85×109/L, hemoglobin ≥ 90g/L;
   2. serum creatinine ≤ 1.5×ULN, creatinine clearance rate ≥60 mL/min, U-pro < 2+ or 1.0g/L; if U-pro ≥2+ or 1.0g/L, 24 hours U-pro ≤ 1.0g/L can be included;
   3. total bilirubin ≤ 1.5×ULN, obstructive jaundice with biliary drainage: total bilirubin ≤ 2.0×ULN; alanine transaminase and aspartate aminotransferase ≤ 2.5×ULN, liver metastasis ≤ 5.0×ULN; serum albumin ≥ 30g/L;
10. Without a history of allergy or hypersensitivity to camptothecin drugs;
11. Taking drugs orally;
12. Serum human chorionic gonadotropin negative in premenopausal women; female patients of childbearing potential and male patients with female partners of childbearing potential must be willing to avoid pregnancy;
13. Ability to understand the study and sign informed consent.

Key exclusion Criteria:

1. Patients who have been previously treated with camptothecin drugs or topoisomerase I inhibitor within 6 months before enrollment;
2. Patients who have been previously treated with gemcitabine and fluorouracil in first-line treatment within 6 months before enrollment;
3. Patients who have been previously treated with other investigational drugs within 4 weeks before enrollment;
4. Patients with brain or meningeal metastasis;
5. Patients with a history of gastrointestinal disease which affects drug absorption;
6. Patients with serous cavity effusion with clinical symptoms (such as pleural effusion, peritoneal effusion, pericardial effusion, etc.), which continue to increase after two-week conservative treatment (excluding puncture drainage);
7. Patients with hypertension that cannot be controlled by drugs (≥ 160/100mmhg); angina pectoris within 3 months before enrollment or unstable angina pectoris; myocardial infarction within 1 year before enrollment and cardiac insufficiency (NYHA ≥ II);
8. Patients with active infections requiring systemic treatment or pyrexia of unknown origin prior to initial administration (except neoplastic fever);
9. Patients with hepatitis B surface antigen positive and peripheral blood hepatitis B virus DNA ≥1.0×103 copy/mL; positive of hepatitis C antibody and peripheral blood hepatitis C virus RNA;
10. Patients with active pulmonary tuberculosis or uncontrolled pulmonary tuberculosis after anti-tuberculosis treatment;
11. Patients with a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases;
12. Patients with a history of malignancies other than pancreatic cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or malignant tumors that have been cured for 5 years;
13. Pregnant or lactating women;
14. Patients with a history of mental diseases (including epilepsy or dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year progression free survival of the whole group.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death from any cause or the date of last follow-up whichever came first, assessed up to 24 months.
  The 2-year overall survival of the whole group.
Objective response rate (ORR) | To evaluate objective response rate every 6 weeks after the initiation of chemotherapy, up to 24 months.
  Percentage of patients with objective response assessed by best overall.
Duration of Response (DoR) | First documented CR or PR, whichever is first recorded until the first assessment of PD, assessed up to 24 months.
  The duration is measured from the first documented response (CR or PR, whichever is first recorded) until the first assessment of Progressive Disease (PD).
Disease control rate (DCR) | To evaluate disease control rate every 6 weeks after the initiation of chemotherapy, up to 24 months.
  Percentage of patients with disease control as assessed by best overall.
Patient-reported outcome (PRO) | To evaluate every 6 weeks after the initiation of chemotherapy, up to 24 months.
  Change from baseline assessed according to the quality of life questionnaire C30.

CONTACTS AND LOCATIONS:
Overall Officials: WANG LIWEI, MD, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Sessa C, Cresta S, Cerny T, Baselga J, Rota Caremoli E, Malossi A, Hess D, Trigo J, Zucchetti M, D'Incalci M, Zaniboni A, Capri G, Gatti B, Carminati P, Zanna C, Marsoni S, Gianni L. Concerted escalation of dose and dosing duration in a phase I study of the oral camptothecin gimatecan (ST1481) in patients with advanced solid tumors. Ann Oncol. 2007 Mar;18(3):561-8. doi: 10.1093/annonc/mdl418. Epub 2006 Dec 5. PMID 17150998
- [Background] Hu J, Wen PY, Abrey LE, Fadul CE, Drappatz J, Salem N, Supko JG, Hochberg F. A phase II trial of oral gimatecan for recurrent glioblastoma. J Neurooncol. 2013 Feb;111(3):347-53. doi: 10.1007/s11060-012-1023-0. Epub 2012 Dec 12. PMID 23232808
- [Background] Pecorelli S, Ray-Coquard I, Tredan O, Colombo N, Parma G, Tisi G, Katsaros D, Lhomme C, Lissoni AA, Vermorken JB, du Bois A, Poveda A, Frigerio L, Barbieri P, Carminati P, Brienza S, Guastalla JP. Phase II of oral gimatecan in patients with recurrent epithelial ovarian, fallopian tube or peritoneal cancer, previously treated with platinum and taxanes. Ann Oncol. 2010 Apr;21(4):759-765. doi: 10.1093/annonc/mdp514. Epub 2009 Nov 11. PMID 19906760